CLINICAL TRIAL: NCT07071220
Title: The Efficacy of Vitamin C Supplementation on Serum IL-6 Levels and Disease Activity in Systemic Lupus Erythematosus Patients
Brief Title: Efficacy of Vitamin C Supplementation on Serum IL-6 Levels and Disease Activity in Systemic Lupus Erythematosus Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sriwijaya (Other)
Responsible Party: Principal Investigator, Yuniza, Principal investigator, Division of Allergy Immunology Faculty Member, Department of Internal Medicine, Universitas Sriwijaya/Mohammad Hoesin General Hospital, Universitas Sriwijaya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04.03/DXVIII0608ETIK/237/2024
Record Dates: First submitted 2025-07-01; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: systemic lupus erythematosus; SLE; vitamin C; IL-6; Mex-SLEDAI; disease activity
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: The study was The study was designed as a single-center double-blind randomized controlled clinical trial. Participants were randomized into two groups receiving Vitamin C or placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple (Participant, Care Provider, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C (Experimental): The patients were given a tablet containing Vitamin C 500 mg twice a day
  Interventions: Dietary Supplement: Vitamin C
- Placebo (Placebo Comparator): The patients were given a placebo capsule with a similar color, shape, size and taste twice a day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C — The patients received vitamin C supplementation
  Arms: Vitamin C
Dietary Supplement: Placebo — Patients received placebo capsules
  Arms: Placebo

SUMMARY:
The study aimed to evaluate the efficacy of vitamin C supplementation compared to placebo towards IL-6 levels and disease activity with the MEX-SLEDAI score in Systemic Lupus Erythematosus (SLE) patients. The current study was designed as a single-center double-blind randomized controlled clinical trial. The participants were voluntarily recruited ≥ 18 years old SLE patients, with mild to moderate disease activity and did not consumed vitamin C 1 week prior to the trial study. Participants were randomized into two groups receiving vitamin C supplementation, or placebo. IL-6 levels and MEX-SLEDAI score were evaluated at the beginning and at the end of the 8 week trial for analysis.

DETAILED DESCRIPTION:
This research is a double blind randomized controlled trial study. The study subjects were 38 patients diagnosed with mild to moderate lupus activity, randomly divided into 2 groups, who received vitamin C supplementation twice daily for 8 weeks and the group that received placebo. Serum IL-6 and the degree of disease activity using MEX-SLEDAI score were measured before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. All patients diagnosed with systemic lupus erythematosus with mild-moderate disease activity who are treated at the Allergy-Immunology Department of RSMH.
2. Patients aged over 18 years.
3. Willing to participate in the study by signing an informed consent form.

Exclusion Criteria

1. Patients with other immune disorders, both autoimmune and immunocompromised conditions such as human immunodeficiency virus (HIV)
2. Pregnant and breastfeeding patients.
3. Patients with malignancies.
4. Patients with chronic liver disorders.
5. Patients with infectious diseases.
6. Patients who consume supplements containing vitamin C.

Drop-out Criteria

1. Patients who discontinue vitamin C for more than 3 weeks.
2. Death.
3. Development of serious drug side effects, requiring discontinuation of the medication.
4. Patients who are readmitted or experience symptom deterioration during the intervention period.
5. Loss to follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
IL-6 | From enrollment to the end of the treatment at 8 weeks
  To determine the effectiveness of adding vitamin C compared to placebo towards IL-6 levels concentration change in SLE patients.
MEX-SLEDAI | From enrollment to the end of the treatment at 8 weeks
  To determine the effectiveness of adding vitamin C compared to placebo towards disease activity in SLE patients, measured with MEX-SLEDAI score

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammad Hoesin General Hospital, Palembang, South Sumatera, Indonesia

REFERENCES:
- [Background] Minami Y, Sasaki T, Arai Y, Kurisu Y, Hisamichi S. Diet and systemic lupus erythematosus: a 4 year prospective study of Japanese patients. J Rheumatol. 2003 Apr;30(4):747-54. PMID 12672194
- [Background] Tam LS, Li EK, Leung VY, Griffith JF, Benzie IF, Lim PL, Whitney B, Lee VW, Lee KK, Thomas GN, Tomlinson B. Effects of vitamins C and E on oxidative stress markers and endothelial function in patients with systemic lupus erythematosus: a double blind, placebo controlled pilot study. J Rheumatol. 2005 Feb;32(2):275-82. PMID 15693087
- [Background] Ellulu MS, Rahmat A, Patimah I, Khaza'ai H, Abed Y. Effect of vitamin C on inflammation and metabolic markers in hypertensive and/or diabetic obese adults: a randomized controlled trial. Drug Des Devel Ther. 2015 Jul 1;9:3405-12. doi: 10.2147/DDDT.S83144. eCollection 2015. PMID 26170625